CLINICAL TRIAL: NCT00131365
Title: Post Approval Study: MR Guided Focused Ultrasound Surgery in the Treatment of Uterine Fibroids
Brief Title: Magnetic Resonance (MR) Guided Focused Ultrasound Surgery of Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF014 - 4.1/3T
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Leiomyoma
Keywords: fibroids; Uterine Fibroids; ExAblate; MrgFUS
MeSH Terms: conditions — Leiomyoma

ARMS (1):
- ExAblate MRgFUS (Experimental): Treatment with the ExAblate 2000 system Version 4.1
  Interventions: Device: ExAblate 2000

INTERVENTIONS:
Device: ExAblate 2000

SUMMARY:
The goal of this study is to develop additional long term data to evaluate the safety and effectiveness of this treatment.

Indications for use for this system is: 'The ExAblate is intended to ablate uterine fibroid tissue in pre- or peri-menopausal women with symptomatic uterine fibroids who desire a uterine sparing procedure. Patients must have a uterine size of less than 24 weeks and not seeking treatment for reasons of improving fertility.'

DETAILED DESCRIPTION:
Background

General:

Uterine leiomyoma (fibroids) are the most common neoplasms of the female pelvis. These benign tumors are generally oval in shape, and often highly vascular. On T2 weighted MR imaging exams, or T1 exams with contrast, uterine fibroids are easily identifiable. They occur in 20-25% of women of reproductive age and can cause a variety of problems generally described as either bleeding or mass effects from the fibroid. In general, these symptoms can be classified into two categories:

1. heavy menstrual bleeding, defined as bleeding on heavy days requiring a change of sanitary wear every 2 hours or less, significant clot passage, flooding, substantial prolongation of menstrual periods compared with the patient's prior experience, or anemia.
2. pelvic pain or pressure, heaviness or discomfort, or similar symptoms in the back, flank or leg attributable to the bulk of the fibroid, urinary frequency, increase in nocturia, difficulty voiding or compression of the ureters with hydronephrosis.

Measures of the clinical success of patients who elect treatment of fibroids are generally subjective, and evaluated by the patient in terms of improvement in the initial symptoms that caused her to seek treatment (decrease in pain, bladder or bowel symptoms, or reduction in vaginal bleeding), while experiencing a minimum of co-morbidities from the treatment itself.

ExAblate Device:

The InSightec ExAblate MR guided Focused Ultrasound Surgery (MRgFUS) system is a non-invasive thermal ablation device fully integrated with an MR imaging system and used for the ablation of soft tissue. It has been evaluated in an earlier FDA international, multi-center study and found to be safe and effective for the treatment of uterine fibroids. ExAblate device received FDA approval in October 2004.

Prior Studies:

The ExAblate has been used for the treatment of uterine fibroids in 2 previous IDE protocols.

* Group A: This was the original Pivotal Study Group (IDE G020001 - Protocol UF002). These 109 patients were treated at 3 sites in the US and at 4 sites outside the US. There was a limitation on the allowable treatment volume and only a single treatment was permitted. Original follow-up was planned for 6 months. The study was later extended to include follow-up visits at 12, 24, and 36 months (UF009). Because of the gap between the initial study consent, and the re-consent for the long term follow-up there was a high dropout rate at the 12 month visit. Thirty-three US patients returned for the 12 months visit, and will continue to be followed for the 24 and 36 M visits.
* Group B: This was the Continued Access Study (IDE G020001 - Protocol UF005) where approximately 160 patients were treated at 3 sites in the US during the PMA review period. Treatment conditions were modified somewhat from the pivotal, including the addition of a second treatment session where necessary. The initial study was planned to include a long term follow-up of 12, 24 and 36 months (UF009).
* Group C: This group of 70 patients (UF14) will be treated post-PMA approval following the commercial treatment guidelines. The follow-up will include for visits at 12, 24 and 36 months. This group includes also another 20 patients who will be treated under this original IDE to validate the ExAblate system for use in a 3T MR scanner, as well as validating a new application SW (V4.1).

ELIGIBILITY:
Inclusion Criteria:

* Women who present with symptomatic uterine fibroids and are not seeking treatment for the reason of improving fertility.
* Able and willing to give consent and able to attend all study visits.
* Patient is pre or peri-menopausal (within 12 months of last menstrual period).
* Able to communicate sensations during the ExAblate procedure.
* Uterine fibroids, which are device accessible (i.e., positioned in the uterus such that they can be accessed without being shielded by bowel or bone).
* Fibroids(s) clearly visible on non-contrast magnetic resonance imaging (MRI).

Exclusion Criteria:

* Metallic implants that are incompatible with MRI
* Sensitive to MRI contrast agents
* Severe claustrophobia that would prevent completion of procedure in MR unit
* Women who are pregnant or desire to become pregnant in the future. Pregnancies following ExAblate treatment could be dangerous for both mother and fetus.
* Pedunculated fibroids
* Active pelvic inflammatory disease (PID)
* Active local or systemic infection
* Known or suspected pelvic carcinoma or pre-malignant conditions, including sarcoma and adenomatous hyperplasia
* Intrauterine device (IUD) anywhere in the treatment path
* Dermoid cyst of the ovary anywhere in the treatment path
* Extensive abdominal scarring that cannot be avoided by redirection of the beam (e.g., due to Caesarean section or repeated abdominal surgeries)
* Undiagnosed vaginal bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Min, M.D., Principal Investigator — Cornell Vascular
Locations (1):
- Cornell Vascular, New York, New York, United States

REFERENCES:
- See also: Sponsor home page — http://www.insightec.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was approved to enroll 20 participants; however, due to the obsolescence of device features the study was closed after enrolling 9 participants.
Period: Overall Study
Arm/Group | ExAblate MRgFUS
Started | 9 (Only safety data was reported due to early closure of the study due to device obsolescence.)
Completed (5 out of 9 enrolled participants were followed through the month 36 visit.) | 5
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Alternative treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | ExAblate MRgFUS
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants] — Age data was not collected
  Participants
    not collected | NA — age data was not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number and Type of Adverse Events
Description: Adverse events outcomes are reported in the adverse events module.
Time Frame: 36 months
Population: Adverse events outcomes are reported in the adverse events module.
Measure: Number; unit: Adverse Events
Groups:
- ExAblate MRgFUS: Treatment with the ExAblate 2000 system Version 4.1
  ExAblate 2000
Arm/Group | ExAblate MRgFUS
Number analyzed (Participants) | 9
Adverse Events | 15

2. Post Hoc Outcome: Number of Subjects With Adverse Events
Description: Adverse events outcomes are reported in the adverse events module.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | ExAblate MRgFUS
Number analyzed (Participants) | 9
Participants | 6

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | ExAblate MRgFUS
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate MRgFUS (N=9)
Abdominal pain (Surgical and medical procedures) | 2 (2)
Discomfort (Surgical and medical procedures) | 2 (2)
Back pain - positional (Surgical and medical procedures) | 1 (1)
Leg/back pain - sonication induced (Surgical and medical procedures) | 1 (1)
Neck pain (Surgical and medical procedures) | 1 (1)
Abdominal pain - sonication related (Surgical and medical procedures) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Foley catheter urethral irritation (Renal and urinary disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 2 (2)
Anal irritation (Gastrointestinal disorders) | 1 (1)
Transient Dysaesthesia (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was closed to enrollment in 2005 due to obsolescence of device features. Only safety data on the 9 enrolled participants was reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No